CLINICAL TRIAL: NCT04038502
Title: An Open-label, Multicenter Phase II Study to Compare the Efficacy of Carboplatin as First-line Followed by Second-line Olaparib Versus Olaparib as First-line Followed by Second-line Carboplatin in the Treatment of Patients With Castration Resistant Prostate Cancer Containing Homologous Recombination Deficiency
Brief Title: Carboplatin or Olaparib for BRcA Deficient Prostate Cancer
Acronym: COBRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ONCA-009-18F; CX-18-006 (Other Grant/Funding Number: Veterans Affairs CSR&D Merit Review Award); 19-08 (Other: VA CIRB); 01783 (Other: MIRB (LSI)); 01781 (Other: MIRB (National Chair)); CX001963-01 (Other: Veterans Affairs CSR&D)
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer; BARD1, BRCA1, BRCA2, BRIP1, CHEK1, FANCL, PALB2; RAD51B, RAD51C, RAD51D, or RAD54L Mutations
Keywords: metastatic prostate cancer
MeSH Terms: conditions — Fanconi Anemia, Complementation Group D1; Hereditary Sensory and Autonomic Neuropathies; Fanconi Anemia, Complementation Group N; Prostatic Neoplasms | interventions — Carboplatin; olaparib

STUDY DESIGN:
Intervention Model Description: Unblinded, randomized (1:1) clinical study with study-drug treatment in metastatic castrate resistant prostate cancer in patients who have inactivation of the homologous DNA repair pathway, including BARD1, BRCA1, BRCA2, BRIP1, CHEK1, FANCL, PALB2, RAD51B, RAD51C, RAD51D, or RAD54L with cross-over to opposite study drug after progression or intolerance (whichever comes first).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm 1 - Carboplatin to Olaparib (Active Comparator): Participants are administered carboplatin AUC 5 IV first, which is administered Cycle-1, Day-1, and then every 21 days as first line therapy. For second line (crossover), olaparib is prescribed and taken orally at home, twice daily, 300 mg in 28 day cycles.
  Interventions: Drug: Carboplatin; Drug: Olaparib
- Treatment Arm 2 - Olaparib to Carboplatin (Active Comparator): Participants are prescribed olaparib which is taken orally at home, twice daily, 300 mg in 28 day cycles, as first line therapy. For second line (crossover), carboplatin is administered AUC 5 IV every 21 days thereafter.
  Interventions: Drug: Carboplatin; Drug: Olaparib

INTERVENTIONS:
Drug: Carboplatin — Chemotherapy FDA approved drug used to treat: ovarian, lung, head and neck cancers. It is sometimes used in combination with other medications or off-label use to treat other metastatic cancers.
  Other Names: Paraplatin
Drug: Olaparib — Olaparib is a targeted therapy drug that is used for mCRPC and is approved by the FDA for this use.
  Other Names: Lynparza

SUMMARY:
This is an unblinded, randomized clinical study comparing the efficacy of DNA damaging chemotherapy using carboplatin, to standard of care therapy for patients who have metastatic castrate resistant prostate cancer. This trial will use olaparib or carboplatin as initial therapy with crossover to the alternate or second-line drug after first progression for patients with tumors containing BARD1, BRCA1, BRCA2, BRIP1, CHEK1, FANCL, PALB2, RAD51B, RAD51C, RAD51D, or RAD54L inactivating mutations.

Participants are randomized (1:1) and receive either carboplatin (AUC 5, IV) every 21 days, first or olaparib taken orally (300 mg), twice daily in 28 day cycles, until intolerance, complete response, or progression by Prostate Cancer Working Group 3 (PCWG3) criteria.

Participants then crossover from the first-line therapy to the second-line therapy with the opposite study medication and receive treatment to intolerance or progression (whichever is first). Enrolled participants will be allowed to crossover to second line therapy if they continue to meet initial eligibility criteria, and at least three weeks have elapsed since last administration of either carboplatin or olaparib. Throughout the study, safety and tolerability will be assessed. Progression will be evaluated with bone scan, CT of the abdomen/pelvis, or MRI and PSA as per PCWG3 criteria.

DETAILED DESCRIPTION:
Study General Trial Over-view

This study is designed to help better understand treatment options compared to standard therapies for patients who have targeted DNA repair mutations and metastatic castrate resistant prostate cancer (mCRPC).

Cancer therapies are aimed at finding a way to kill the cancer cells while causing minimal damage to normal (non-cancer) cells. This often works because cancers cells grow faster than many normal cells, many treatments are aimed at to take advantage of that difference. One of the ways to do this is to damage the DNA of these more rapidly growing cells. However, if the cells have a way of repairing that damage then therapies may not work as well. Some research shows that when specific changes or mutations occur in the genes involved with repairing DNA damage, resulting cancers have responded well to drugs which damage DNA.

Olaparib is known as a PARP inhibitor and is standard of care therapy for men with BRCA altered mCRPC. Carboplatin is a synthetic antineoplastic agent which has been used in the treatment of solid tumors and BRCA related cancers. When mutations occur in critical DNA-repair genes, research has found that treatment with carboplatin is also effective.

This research is being done to determine the response of mCRPC in patients with DNA repair mutations to treatment with olaparib compared to carboplatin. This study will test whether giving one drug or the other a has a better response.

Patients wishing to participate in this study are screened for safety and health eligibility before enrolling.

This study is enrolling 100 male participants total, from across the VAMC nationally who have the following:

* Metastatic castration-resistant prostate cancer (mCRPC)
* Cancer that has gotten worse, after any number of first-line treatments
* Mutations in DNA-repair genes discovered as part of a patient's routine care.

Once eligibility is determined, enrolled participants are randomized into one of two groups:

* Group A will start with carboplatin (IV) first, given every 21 days, then have the option to switch to the second treatment with olaparib taken daily, (orally) with cycles of every 28 days.
* Group B will start with olaparib first, taken (orally), with 28 day cycles, then have the option to switch to the second treatment with carboplatin (IV) every 21 days.

Both study drugs in this trial are currently FDA approved, and are prescribed at the participating VAMC clinical sites per institutional guidelines. Carboplatin given in IV is also given as prescribed at the participating VAMC, and administered per institutional guidelines.

Participants are monitored for health and body function, cancer progression, toxicity and life quality at every visit during the trial and at an end of treatment visit (28 days after completion of the trial or after withdrawal). For participants who respond well to treatment during the trial, additional treatment cycles may be added and the study can be extended. Participants who experience intolerable toxicity, cancer progression, or whose doctors decide to change treatment, will either be switched to the opposite study drug or withdrawn from the study.

This important trial is designed to compare response rate and duration of response using carboplatin compared to olaparib in patients who have mCRPC which contains DNA repair gene mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Signed study informed consent form (ICF) and HIPAA authorization form
2. Male age > 18 years
3. Diagnosis of prostate cancer (pure small-cell histology or pure high-grade neuroendocrine histology are excluded; neuroendocrine differentiation is allowed)
4. Ongoing gonadal androgen deprivation therapy with gonadotropin-releasing hormone (GnRH) analogues, antagonists or orchiectomy. Patients who have not had an orchiectomy must be maintained on effective GnRH analogue/antagonist therapy
5. mCRPC as defined by serum testosterone < 50 ng/ml (for patients on GnRH analogues or antagonists) and at least one of the following:

   * PSA level of at least 2 ng/ml that has risen on at least 2 successive occasions at least 1 week apart
   * Evaluable disease progression by modified RECIST 1.1 (Response Evaluation Criteria in Solid Tumors)
   * Progression of metastatic bone disease on bone scan, CT or MRI with > 2 new lesions
6. Prior therapy with abiraterone acetate, enzalutamide, apalutamide, or darolutamide
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of < 2 (see Appendix 3, ECOG Grading Scale)
8. Results of previous standard DNA testing, or previous research testing, which confirms RAD51B, RAD51C, RAD51D, or RAD54L mutations (see Introduction, Section 2 for study design and previous research on targeted therapy) from primary, metastatic tumor or circulating tumor DNA, or pathogenic/likely pathogenic germline variant as assessed by a CLIA certified laboratory level assay for DNA sequencing.
9. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   * Hemoglobin > 10.0 g/dL
   * Absolute neutrophil count (ANC) > 1.5 x 109/L
   * Platelet count > 100 x 109/L
   * Total bilirubin < 1.5 x institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) < 2.5 x institutional upper limit of normal unless liver metastases are present in which case, they must be < 5x ULN
   * Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of >51 mL/min: Estimated creatinine clearance =(140-age [years]) x weight (kg))/ (serum creatinine (mg/dL) x 72)

Exclusion Criteria:

1. Currently receiving active therapy for other neoplastic disorder(s)
2. Concurrent enrollment in another clinical investigational drug or device study
3. Histologic evidence of small cell carcinoma (morphology alone - immunohistochemical evidence of neuroendocrine differentiation without morphologic evidence is not exclusionary)
4. Prior treatment with platinum, mitoxantrone or PARP inhibitor for castration resistant prostate cancer
5. Known parenchymal brain metastasis
6. Active or symptomatic viral hepatitis or chronic liver disease AST or ALT > 2.5 x ULN or total bilirubin > ULN (unless Gilbert's syndrome is the etiology of hyperbilirubinemia)
7. Subjects with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML
8. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks
9. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for phenobarbital and 3 weeks for other agents
10. Subjects unable to swallow orally administered medication and subjects with gastrointestinal disorders likely to interfere with absorption of the study medication
11. Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 35 % at baseline
12. Treatment with an investigational therapeutic within 30 days of Cycle-1
13. Presence of dementia, psychiatric illness, and/or social situations limiting compliance with study requirements or understanding HIPAA authorization and/or giving of informed consent
14. Any condition(s), medical or otherwise, which, in the opinion of the Investigators, would jeopardize either the patient or the integrity of the data obtained.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically sexed males with metastatic prostate cancer
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS-1L) defined as the time interval between randomization and first documented disease progression or death due to any cause reported during, or after, first-line treatment. | Through duration of the study, up to six years
  Progression free survival (PFS) by bone scan or measurable disease, Response Evaluation Criteria in Solid Tumors (RECIST 1.1) to initial therapy (PFS-1L) with either study drug.

SECONDARY OUTCOMES:
time interval between randomization and second documented disease progression during or after second-line or death (due to any cause) | Through duration of the study, up to six years
  Progression-free survival combined, a composite endpoint defined as the time interval between randomization and second documented disease progression reported during or after second-line or death due to any cause
PSA measurements/response | Through duration of the study, up to six years
  To assess PSA response to initial therapy with carboplatin vs. olaparib
PSA measurements/response | Through duration of the study, up to six years
  To assess PSA response duration to second line therapy with olaparib vs carboplatin
Grade 3 and 4 toxicities in first and second-line setting | Through duration of the study, up to six years
  To assess Grade 3 and 4 toxicities for each regimen in the first- and second-line setting

OTHER OUTCOMES:
Exploratory Objective - PFS | Through duration of the study, up to six years
  To assess the PFS of patients who receive olaparib versus patients who receive carboplatin during the second-line of treatment (PFS-2L)
Exploratory Objective - objective response rate | Through duration of the study, up to six years
  To assess the objective response rate in patients who receive olaparib versus patients who receive carboplatin during second-line of treatment.
Exploratory Objective- objective duration of response | Through duration of the study, up to six years
  To assess the objective duration of response in patients who receive olaparib versus patients who receive carboplatin during second-line of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. Montgomery, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Ryan Burri, MD, Principal Investigator — Bay Pines VA Healthcare System, Pay Pines, FL; Phoebe Tsao, MD MSc, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Maneesh Jain, MD, Principal Investigator — Washington DC VA Medical Center, Washington, DC
Locations (18):
- United States (18):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Boise VA Medical Center, Boise, ID, Boise, Idaho
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Philadelphia MultiService Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No